CLINICAL TRIAL: NCT02132026
Title: SALTIRE II: Bisphosphonates and RANKL Inhibition in Aortic Stenosis
Brief Title: Study Investigating the Effect of Drugs Used to Treat Osteoporosis on the Progression of Calcific Aortic Stenosis.
Acronym: SALTIRE II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other); NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SALTIRE2-2014
Record Dates: First submitted 2014-05-02; First posted 2014-05-06 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2020-03

CONDITIONS: Calcific Aortic Stenosis
Keywords: Aortic Stenosis; Denosumab; Alendronic Acid; Osteoporosis
MeSH Terms: conditions — Aortic Valve, Calcification of; Aortic Valve Stenosis; Osteoporosis | interventions — Denosumab; Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alendronic Acid (Active Comparator): 50 patients will receive once weekly Alendronic Acid tablets (70mg).
  Interventions: Drug: Alendronic Acid
- Alendronic Acid placebo (Placebo Comparator): 25 patients will receive alendronic acid placebo tablets.
  Interventions: Drug: Alendronic Acid Placebo
- Denosumab (Active Comparator): 50 patients will receive 6 monthly denosumab injections
  Interventions: Drug: Denosumab
- Denosumab Placebo (Placebo Comparator): 25 patients will receive a 6 monthly placebo injection.
  Interventions: Drug: Denosumab Placebo

INTERVENTIONS:
Drug: Denosumab
  Other Names: Prolia; Marketing Authorisation Number : EU/1/11/703/003; ATC number M05BX04
  Arms: Denosumab
Drug: Alendronic Acid
  Other Names: Marketing Authorisation Number PL 30306/0032; ATC codes M05B A04
  Arms: Alendronic Acid
Drug: Denosumab Placebo — subcutaneous injection of 0.9%Saline at baseline, 6 months, 12 months and 18 months
  Arms: Denosumab Placebo
Drug: Alendronic Acid Placebo — Inert Capsule containing lactose monohydrate manufactured and labelled by Investigational Supplies Group (ISG) University of Edinburgh.
  Arms: Alendronic Acid placebo

SUMMARY:
Aortic stenosis is a condition whereby one of the heart valves (aortic valve) becomes narrowed, due to calcium deposition, over time. This can lead to chest pain, heart failure and sudden death. It is the commonest valve disease requiring surgery in the developed world and as the population becomes increasingly older, it is predicted that the prevalence of aortic stenosis will double in the next 20 years. Currently the only treatment is replacement of the aortic valve. Whilst this is excellent treatment, not everyone is suitable for it.

The primary objective of our study is to determine whether 2 drugs used in the treatment of osteoporosis (a condition of bone thinning) can halt/retard the progression of aortic stenosis. This is on the basis that studies have suggested that altered regulation of calcium metabolism may be an important mechanism perpetuating the disease. Both drugs work by reducing calcium release into the bloodstream from bones and therefore calcification of the aortic valve.

150 patients will therefore be randomly allocated to either of the trial drugs which are denosumab,the bisphosphonate (alendronic acid), or a placebo.

Positron Emission Tomography (PET) scanning is a technique where biochemically active molecules are injected and are taken up at sites of ongoing calcification activity where they emit radiation and can be detected by the PET scanner. We have previously shown that this technique can demonstrate areas of newly developing calcification on an aortic valve.

We therefore propose that patients receiving bisphosphonates or denosumab will have reduced evidence of active calcification and slower progression of their disease at two years as assessed by Echocardiography (ultrasound) and a change in their calcium score (quantity of calcium on the aortic valve measured using Computed Tomography [CT] ).

The data from this study will then be used to design a larger trial.

DETAILED DESCRIPTION:
BACKGROUND Aortic Stenosis is a common cause of valvular heart disease in which the valve cusps become progressively calcified. The only available treatment is aortic valve replacement and previous attempts at providing medical therapies to modify the disease process have proved unsuccessful.

Pathophysiology of Aortic Stenosis. The initiating event is believed to be caused by mechanical damage to the cells lining the valve in a process similar to that which occurs in atherosclerosis. However the propagating mechanism is more likely to be that of active calcification. In support of this, a growing body of pre-clinical and clinical data indicates that treatments for osteoporosis, which work by preventing the breakdown of bone and therefore calcium release into the blood, can reduce calcium deposition (calcification) of the blood vessels. These agents therefore hold considerable promise as novel therapies for aortic stenosis.

Denosumab in Aortic Stenosis Denosumab is a drug which prevents bone cells called osteoclasts from breaking down bone and releasing calcium into the blood. For this reason it is used to treat osteoporosis. It works on a specific pathway which we believe to be important in regulating calcium release from bone. Mice engineered with defects within this pathway were found to have increased bone breakdown and blood vessel calcification. Furthermore there have been two studies to assess the role of this pathway in patients with aortic valve disease. Both studies have also demonstrated altered regulation within this pathway

Bisphosphonates in Aortic Stenosis Bisphosphonates are a group of drugs widely used for the treatment of osteoporosis and also prevent bone breakdown by osteoclasts. They have also been shown to have important cardiovascular effects with a consistent reduction in calcification of blood vessels and the aortic valve. This in part appears to be a consequence of their inhibition of bone breakdown but also by reducing the production of key inflammatory substances implicated in the early stages of aortic stenosis. We plan on using alendronic acid which is a bisphosphonate commonly used in the management of osteoporosis.

PET CT scanning in Aortic Stenosis. 18F-NaF (Sodium Fluoride) is biochemical compound which preferentially binds to regions of newly developing calcification and emits radiation. When used in combination with Computed Tomography (CT) it enables it to be localized. This way we are able to identify areas of newly developing calcification on an aortic valve.

In previous studies in our institution, we demonstrated we could quantify 18F-NaF uptake in the aortic valve and that there was a progressive rise in activity with increasing disease severity. We found that at At 1 year, the baseline 18F-NaF uptake emerged as a powerful predictor of the progression in aortic valve calcification. Following analysis of 2 year follow up data, 18F-NaF emerged as an independent predictor of aortic valve replacement and cardiovascular mortality

Therefore these findings have led us to propose that

1. Calcification is the key driver to Aortic Stenosis Progression
2. We want to reduce calcification activity using Denosumab and Biphosphonates
3. We predict that this will reduce the 18F-NaF signal and disease progression on Echocardiography and CT.

STUDY DESIGN This will be a double-blind, randomized, placebo-control trial of denosumab and alendronic acid in patients with aortic stenosis.

Study population and randomization

We aim to recruit 170 patients in total with non-rheumatic calcific aortic stenosis.

20 patients will only participate in scan-rescan reproducibility studies. They will not proceed to the randomization stage.

Of the remaining 150 patients, 75 subjects will be randomized (2:1) to either subcutaneous denosumab 60 mg (n=50) or matched placebo (n=25) every 6 months; and a further 75 will be randomized (2:1) to oral alendronate 70 mg (n=50) or matched placebo (n=25) once weekly

Assessment and follow up

All subjects will undergo a standardized clinical assessment at baseline and every six months. Data will be collected with respect to symptomatic status, the trial safety endpoints, routine biochemical profiling, biomarkers, quality of life questionnaires and electrocardiography.

Aortic stenosis severity will be assessed at baseline and every 6 months by echocardiography performed by a single, dedicated sonographer to maximize reproducibility. Severity will be assessed using the peak and mean aortic valve pressure gradients (this technique is used to monitor aortic stenosis severity; the higher the pressure gradient across the aortic valve the more severe the narrowing). We will also calculate the aortic valve area and calcification score.

PET CT and CT calcium scoring.

Both will be performed using a combined PET and 128-multidetector CT scanner (Biograph 128, Siemens).

CT calcium scoring measures the amount of calcium in the valve and will be assessed at baseline, 6 months and 2 years. It will act as an additional marker of disease severity and progression alongside Echocardiography. Those with a heart rate of >65 /min will be given heart-slowing medication (beta blockers) if deemed safe. The region of the aortic valve will be then be scanned during a breath hold.

18F-NaF PET uptake will be measured at baseline, and 6 months to assess the early impact of the intervention on valvular calcification activity. PET images on their own are difficult to interpret as they do not tell you where the radiation is coming from. For this reason the PET needs to be performed alongside CT which gives us images of the aortic valve. By superimposing the two images we are able to identify where the 'PET signal' is originating from.

To ensure optimal image quality patients will be required to adhere to a high fat, low carbohydrate diet for 48 hours prior to the scan. The subject will then be cannulated to enable injection of the 18F-NaF tracer. They will then rest in a quiet environment for 60 minutes to enable the tracer to reach the valve before transfer to the imaging suite. Those with a heart rate of >65 /min will be given beta-blockade if it is deemed suitable and safe. This is routine practice in cardiac CT. A scout CT will be performed to allow optimal alignment of the PET and CT scanners (so we can be sure the radiation we are detecting is coming from the aortic valve). The patient will then be asked to lie still for 30 minutes so that the PET data can be acquired.

Finally a 'CT angiogram' will be performed of the aortic valve. This involves image acquisition following injection of a radio opaque dye into the aorta. This again allows more accurate localization of our PET signal.

The additional twenty patients will only undergo repeat PET/CT imaging within 2 weeks of their baseline scan to investigate scan-rescan reproducibility of the 18F-NaF PET signal. They will not proceed with the trial beyond this stage to avoid facing increased radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

1. age >50 years
2. peak aortic jet velocity of >2.5 m/s on Doppler echocardiography
3. grade 2-4 calcification of the aortic valve on echocardiography

Exclusion Criteria:

1. Anticipated or planned aortic valve surgery in the next 6 months,
2. Life expectancy <2 years,
3. Inability to undergo scanning
4. Treatment for osteoporosis with bisphosphonates or denosumab.
5. Long-term corticosteroid use.
6. Abnormalities of the oesophagus or conditions which delay oesophageal/gastric emptying,

8) Inability to sit or stand for at least 30 minutes, 9) Known allergy or intolerance to alendronate or denosumab, or any of their excipients, 10) Hypocalcaemia, 11) Maintenance calcium supplementation, 12) Dental extraction within 6 months, 13) History of osteonecrosis of the jaw, 14) Major or untreated cancers, 15) Poor dental hygiene, 16) Women of child-bearing potential who have experienced menarche, are pre-menopausal, have not been sterilised or who are currently pregnant, 17) Women who are breastfeeding, 18) Renal failure (estimated glomerular filtration rate of <30 mL/min), 19) Allergy or contraindication to iodinated contrast, 20) Inability or unwilling to give informed consent, 21) Likelihood of non-compliance to treatment allocation or study protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-11-12 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Change in aortic valve calcium score | Measured at Baseline, 6 months and 2 years
  The change in calcium score will be assessed using computed tomography and is an assessment of disease severity.

SECONDARY OUTCOMES:
Change in aortic valve 18F-NaF uptake | Measured at baseline and 6 months
  This is determined by positron emission tomography and is a measure of calcification activity.
Change in aortic-jet velocity | Measured at baseline, 6, 12, 18 and 24 months
  This will be determined by Doppler echocardiography and is a measure of disease severity.
Change in thoracic aortic and coronary artery calcium score | Measured at baseline and 2 years
  This will be determined by computed tomography and is an additional assessment of vascular calcification.
Change in thoracic spine bone mineral density | Measured at baseline and 2 years
  This will be determined by quantitative computed tomography.
Change in quality of life determined by Short Form 36 Questionnaire | Measured at baseline and 2 years
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rong Bing, MbChB, Principal Investigator — University of Edinburgh; David E Newby, BA BSc PhD BM DM FRCP DSc FRSE, Study Chair — University of Edinburgh
Locations (1):
- Clinical Research Facility University of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- [Background] Dweck MR, Jenkins WS, Vesey AT, Pringle MA, Chin CW, Malley TS, Cowie WJ, Tsampasian V, Richardson H, Fletcher A, Wallace WA, Pessotto R, van Beek EJ, Boon NA, Rudd JH, Newby DE. 18F-sodium fluoride uptake is a marker of active calcification and disease progression in patients with aortic stenosis. Circ Cardiovasc Imaging. 2014 Mar;7(2):371-8. doi: 10.1161/CIRCIMAGING.113.001508. Epub 2014 Feb 7. PMID 24508669
- [Background] Dweck MR, Khaw HJ, Sng GK, Luo EL, Baird A, Williams MC, Makiello P, Mirsadraee S, Joshi NV, van Beek EJ, Boon NA, Rudd JH, Newby DE. Aortic stenosis, atherosclerosis, and skeletal bone: is there a common link with calcification and inflammation? Eur Heart J. 2013 Jun;34(21):1567-74. doi: 10.1093/eurheartj/eht034. Epub 2013 Feb 7. PMID 23391586
- [Background] Dweck MR, Joshi FR, Newby DE, Rudd JH. Noninvasive imaging in cardiovascular therapy: the promise of coronary arterial (1)(8)F-sodium fluoride uptake as a marker of plaque biology. Expert Rev Cardiovasc Ther. 2012 Sep;10(9):1075-7. doi: 10.1586/erc.12.104. No abstract available. PMID 23098140
- [Background] Dweck MR, Jones C, Joshi NV, Fletcher AM, Richardson H, White A, Marsden M, Pessotto R, Clark JC, Wallace WA, Salter DM, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Assessment of valvular calcification and inflammation by positron emission tomography in patients with aortic stenosis. Circulation. 2012 Jan 3;125(1):76-86. doi: 10.1161/CIRCULATIONAHA.111.051052. Epub 2011 Nov 16. PMID 22090163
- [Derived] Oikonomou EK, Craig NJ, Holste G, Vasisht Shankar S, White A, Mahendran M, Newby DE, Dweck MR, Khera R. Artificial Intelligence-Enabled Echocardiography as a Surrogate for Multimodality Aortic Stenosis Imaging: Post Hoc Analysis of a Clinical Trial. Circ Cardiovasc Imaging. 2025 Dec 31:e018353. doi: 10.1161/CIRCIMAGING.125.018353. Online ahead of print. PMID 41473954
- [Derived] Geers J, Manral N, Razipour A, Park C, Tomasino GF, Xing E, Grodecki K, Kwiecinski J, Pawade T, Doris MK, Bing R, White AC, Droogmans S, Cosyns B, Slomka PJ, Newby DE, Dweck MR, Dey D. Epicardial adipose tissue, myocardial remodelling and adverse outcomes in asymptomatic aortic stenosis: a post hoc analysis of a randomised controlled trial. Heart. 2025 Jun 26;111(14):686-694. doi: 10.1136/heartjnl-2024-324925. PMID 40050004
- [Derived] Geers J, Bing R, Pawade TA, Doris MK, Daghem M, Fletcher AJ, White AC, Forsyth L, Evans E, Kwiecinski J, Williams MC, van Beek EJR, Kwak S, Peeters FECM, Tzolos E, Slomka PJ, Lucatelli C, Ralston SH, Prendergast B, Newby DE, Dweck MR. Effect of Denosumab or Alendronate on Vascular Calcification: Secondary Analysis of SALTIRE2 Randomized Controlled Trial. J Am Heart Assoc. 2024 Sep 17;13(18):e032571. doi: 10.1161/JAHA.123.032571. Epub 2024 Sep 9. PMID 39248270
- [Derived] Pawade TA, Doris MK, Bing R, White AC, Forsyth L, Evans E, Graham C, Williams MC, van Beek EJR, Fletcher A, Adamson PD, Andrews JPM, Cartlidge TRG, Jenkins WSA, Syed M, Fujisawa T, Lucatelli C, Fraser W, Ralston SH, Boon N, Prendergast B, Newby DE, Dweck MR. Effect of Denosumab or Alendronic Acid on the Progression of Aortic Stenosis: A Double-Blind Randomized Controlled Trial. Circulation. 2021 Jun 22;143(25):2418-2427. doi: 10.1161/CIRCULATIONAHA.121.053708. Epub 2021 Apr 29. PMID 33913339
- [Derived] Pawade T, Clavel MA, Tribouilloy C, Dreyfus J, Mathieu T, Tastet L, Renard C, Gun M, Jenkins WSA, Macron L, Sechrist JW, Lacomis JM, Nguyen V, Galian Gay L, Cuellar Calabria H, Ntalas I, Cartlidge TRG, Prendergast B, Rajani R, Evangelista A, Cavalcante JL, Newby DE, Pibarot P, Messika Zeitoun D, Dweck MR. Computed Tomography Aortic Valve Calcium Scoring in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2018 Mar;11(3):e007146. doi: 10.1161/CIRCIMAGING.117.007146. PMID 29555836
- [Derived] Pawade TA, Cartlidge TR, Jenkins WS, Adamson PD, Robson P, Lucatelli C, Van Beek EJ, Prendergast B, Denison AR, Forsyth L, Rudd JH, Fayad ZA, Fletcher A, Tuck S, Newby DE, Dweck MR. Optimization and Reproducibility of Aortic Valve 18F-Fluoride Positron Emission Tomography in Patients With Aortic Stenosis. Circ Cardiovasc Imaging. 2016 Oct;9(10):e005131. doi: 10.1161/CIRCIMAGING.116.005131. PMID 27733431
- [Derived] Pawade TA, Newby DE, Dweck MR. Calcification in Aortic Stenosis: The Skeleton Key. J Am Coll Cardiol. 2015 Aug 4;66(5):561-77. doi: 10.1016/j.jacc.2015.05.066. PMID 26227196
- [Derived] Pawade TA, Newby DE. Treating aortic stenosis: arresting the snowball effect. Expert Rev Cardiovasc Ther. 2015 May;13(5):461-3. doi: 10.1586/14779072.2015.1037284. Epub 2015 Apr 16. PMID 25882205